CLINICAL TRIAL: NCT04359940
Title: The Effect of Different Contouring Techniques on Cardiac Magnetic Resonance Assessment of Right Ventricular Volumes in Repaired Tetraology of Fallot: Implications on Preoperative Thresholds for Intervention
Brief Title: Effect of Contouring Techniques on CMR Assessment of the Right Ventricle in Repaired Tetraology of Fallot
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, William E Moody, Consultant Cardiologist, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: CARMS
Record Dates: First submitted 2020-04-13; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Tetralogy of Fallot
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Repaired Tetralogy of Fallot: Patients undergoing routine clinical aand CMR surveillance
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — For clinical surveillance

SUMMARY:
Patients with repaired tetralogy of Fallot (RTOF) develop chronic pulmonary regurgitation and require monitoring for right ventricular dilatation. Pulmonary valve replacement can prevent irreversible right ventricular (RV) dilatation and dysfunction and cardiac magnetic resonance (CMR) is used to facilitate its optimal timing. The investigators sought to determine whether the choice of myocardial contouring technique affects preoperative RV volumetric thresholds for intervention.

DETAILED DESCRIPTION:
Participants with repaired tetralogy of Fallot (RTOF) will be identified using existing patient electronic records who have developed chronic pulmonary regurgitation and are undergoing monitoring for right ventricular dilatation. Cardiac magnetic resonance (CMR) is used to facilitate its optimal timing. Pulmonary valve replacement can prevent irreversible right ventricular (RV) dilatation and dysfunction and cardiac magnetic resonance (CMR) is used to facilitate its optimal timing. There are different post-processing techniques published for measuring RV volumes on cardiac magnetic resonance imaging (detailed vs. smoothed and manual vs. automated). The primary aim of this study is to identify whether the choice of myocardial contouring technique affects the preoperative RV volumetric thresholds for intervention. As a secondary aim, the investigators will determine the reproducibility of different contouring methods.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with repaired Tetralogy of Fallot undergoing routine clinical surveillance at a Level 1 ACHD surgical referral centre.

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with repaired tetralogy of Fallot (RTOF) with chronic pulmonary regurgitation who require monitoring for right ventricular dilatation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Estimated)

PRIMARY OUTCOMES:
Difference in the baseline measurement of indexed right ventricular end-diastolic volume according to the contouring technique | Cross-sectional study. Repeated measurements performed on the baseline CMR study.
  Measurements of indexed right ventricular end-diastolic volume will be repeated using different contouring techniques on the same cardiac MRI study performed at baseline pre-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: William Moody, Principal Investigator — UHB
Locations (2):
- United Kingdom (2):
  - QEHB, Birmingham
  - Cardiac MRI department, University Hospitals Birmingham NHS Foundation Trust, Birmingham

IPD SHARING:
Plan to Share IPD: No